CLINICAL TRIAL: NCT01922336
Title: A Randomised, Single-blind, Three-arm, Parallel Group, Single-dose Study to Compare the Pharmacokinetics, Safety, Tolerability, and Immunogenicity of Three Formulations of Infliximab (SB2, EU Sourced Remicade® and US Sourced Remicade®) in Healthy Subjects
Brief Title: Pharmacokinetic, Safety, Tolerability and Immunogenicity Study of SB2 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Samsung Bioepis Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: SB2-G11-NHV; 2012-005306-22 (EudraCT Number)
Record Dates: First submitted 2013-08-12; First posted 2013-08-14 (Estimated); Results first posted 2019-02-21 (Actual); Last update posted 2019-02-21 (Actual); Status verified 2018-10

CONDITIONS: Healthy
Keywords: Pharmacokinetics

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- SB2 (Experimental): SB2 (Study drug)
  Interventions: Biological: SB2
- EU Remicade (Active Comparator): EU sourced Remicade (Reference drug)
  Interventions: Biological: EU Remicade
- US Remicade (Active Comparator): US sourced Remicade (Reference drug)
  Interventions: Biological: US Remicade

INTERVENTIONS:
Biological: SB2 — IV infusion
  Arms: SB2
Biological: EU Remicade — IV infusion
  Arms: EU Remicade
Biological: US Remicade — IV infusion
  Arms: US Remicade

SUMMARY:
The purpose of this study is to compare the pharmacokinetics, safety, tolerability and immunogenicity of SB2 and Remicade (EU sourced Remicade and US sourced Remicade) in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female subjects of non-childbearing potential and healthy male subjects
* Have a body weight between 60.0 and 94.9 kg and a body mass index between 20.0 and 29.9 kg/m², inclusive.

Exclusion Criteria:

* history and/or current presence of clinical significant atopic allergy, hypersensitivity or allergic reactions, also including known or suspected clinically relevant drug hypersensitivity to any components of the test and reference IP formulation or comparable drugs.
* active or latent Tuberculosis or who have a history of Tuberculosis.
* history of invasive systemic fungal infections or other opportunistic infections
* systemic or local infection, a known risk for developing sepsis and/or known active inflammatory process
* serious infection associated with hospitalisation and/or which required intravenous antibiotics
* history of and/or current cardiac disease
* have received live vaccine(s) within 30 days prior to Screening or who will require live vaccine(s) between Screening and the final study visit.
* Intake medication with a half-life > 24 h within 1 month or 10 half-lives of the medication prior to the administration of investigational product.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 159 (Actual)
Dates: Start 2013-07; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rainard Fuhr, M.D., Ph.D., Principal Investigator — Parexel
Locations (1):
- Parexel International GmbH, Berlin, Germany

REFERENCES:
- [Derived] Shin D, Kim Y, Kim YS, Kornicke T, Fuhr R. A Randomized, Phase I Pharmacokinetic Study Comparing SB2 and Infliximab Reference Product (Remicade((R))) in Healthy Subjects. BioDrugs. 2015 Dec;29(6):381-8. doi: 10.1007/s40259-015-0150-5. PMID 26577771

RESULTS

PARTICIPANT FLOW:
Groups:
- SB2 (Proposed Infliximab Biosimilar): SB2 (Study drug)
  SB2: IV infusion
Period: Overall Study
Arm/Group | SB2 (Proposed Infliximab Biosimilar) | EU Remicade | US Remicade
Started | 53 | 53 | 53
Completed | 53 | 53 | 53
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SB2 (Proposed Infliximab Biosimilar) | EU Remicade | US Remicade | Total
Number analyzed (Participants) | 53 | 53 | 53 | 159
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.7 (9.67) | 40.3 (9.72) | 39.4 (9.87) | 40.1 (9.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 3 | 9
  Male | 49 | 51 | 50 | 150
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 51 | 52 | 52 | 155
  Asian | 1 | 0 | 1 | 2
  Black or African American | 1 | 0 | 0 | 1
  Other | 0 | 1 | 0 | 1
BMI [Mean (Standard Deviation); unit: kg/m2] | 24.56 (2.078) | 25.39 (2.092) | 24.79 (2.058) | 24.91 (2.092)

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve From Time Zero to Infinity (AUCinf)
Time Frame: 71 days
Measure: Mean (Standard Deviation); unit: h·μg/mL
Arm/Group | SB2 (Proposed Infliximab Biosimilar) | EU Remicade | US Remicade
Number analyzed (Participants) | 51 | 53 | 53
h·μg/mL | 38702.8145 (11113.62172) | 39359.7493 (12332.41615) | 39270.1707 (10064.08853)

2. Primary Outcome: Maximum Serum Concentration (Cmax)
Time Frame: 71 days
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | SB2 (Proposed Infliximab Biosimilar) | EU Remicade | US Remicade
Number analyzed (Participants) | 51 | 53 | 53
μg/mL | 126.9975 (16.89586) | 126.2377 (17.88151) | 129.1508 (18.75573)

3. Primary Outcome: Area Under the Concentration-time Curve From Time Zero to the Last Quantifiable Concentration (AUClast)
Time Frame: 71 days
Measure: Mean (Standard Deviation); unit: h·μg/mL
Arm/Group | SB2 (Proposed Infliximab Biosimilar) | EU Remicade | US Remicade
Number analyzed (Participants) | 51 | 53 | 53
h·μg/mL | 36862.4180 (9132.75342) | 37022.3524 (9398.42182) | 37367.5577 (8332.05331)

4. Secondary Outcome: Time to Cmax (Tmax)
Time Frame: 71 days
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | SB2 (Proposed Infliximab Biosimilar) | EU Remicade | US Remicade
Number analyzed (Participants) | 51 | 53 | 53
hour | 2.9294 (1.11529) | 2.5824 (0.95950) | 2.7591 (1.03184)

ADVERSE EVENTS:
Arm/Group | SB2 (Proposed Infliximab Biosimilar) | EU Remicade | US Remicade
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/53 | 0/53
Serious Adverse Events (participants affected / at risk) | 2/53 | 0/53 | 0/53
Other Adverse Events (participants affected / at risk) | 14/53 | 11/53 | 13/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SB2 (Proposed Infliximab Biosimilar) (N=53) | EU Remicade (N=53) | US Remicade (N=53)
Borrelia infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Renal cyst ruptured (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SB2 (Proposed Infliximab Biosimilar) (N=53) | EU Remicade (N=53) | US Remicade (N=53)
Nasopharyngitis (Infections and infestations) | 6 (6) | 4 (4) | 13 (13)
Headache (Nervous system disorders) | 5 (9) | 6 (8) | 7 (7)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 2 (2) | 1 (1)
Rhinitis (Infections and infestations) | 3 (3) | 2 (2) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes